CLINICAL TRIAL: NCT03647124
Title: A Non-interventional, Post-authorization Safety Study of Patients With Relapsed or Refractory Mantle Cell Lymphoma to Further Investigate and Characterize the Association of Lenalidomide With Tumor Flare Reaction and High Tumor Burden
Brief Title: A Study to Evaluate the Relationship of Lenalidomide With Tumor Flare Reaction and High Tumor Burden in Participants With Relapsed or Refractory Mantle Cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-5013-MCL-005; U1111-1213-1816 (Registry Identifier: WHO); EUPAS23366 (Registry Identifier: EU PAS Register)
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Lymphoma, Mantle-Cell
Keywords: Mantle Cell Lymphoma; MCL; Revlimid; Non-Interventional; PASS; CC-5013; Relapsed; Refractory; TFR; Tumor Flare Reaction; High Tumor Burden
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Recurrence | interventions — Lenalidomide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lenalidomide treated Relapsed or refractory mantle cell lymphoma (R/R-MCL) participants in Europe
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Specified dose on specified days
  Other Names: Revlimid; L04AX04

SUMMARY:
The purpose of this study is to investigate and characterize the association of lenalidomide with tumor flare reaction and high tumor burden in participants with relapsed or refractory mantle cell lymphoma.

DETAILED DESCRIPTION:
This is a European multinational, retrospective, non-interventional study of participants with relapsed or refractory mantle cell lymphoma (R/R MCL). Potential sites will be identified where R/R MCL participants have been treated with lenalidomide. Site inclusion will be limited to countries where lenalidomide is reimbursed for this indication.

ELIGIBILITY:
Inclusion Criteria:

Received at least one dose of lenalidomide commencing after 08 July 2016 for the treatment of relapsed refractory mantle cell lymphoma.

Informed consent of the patient or an authorized third person or authority, if required by law, given prior to data collection.

Patient must be ≥18 years of age at the time of signing the informed consent form.

Exclusion Criteria:

1) Patients will be excluded if they were participating in an interventional clinical trial during the treatment period under observation in this Post Authorization Safety Study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of a retrospective cohort of participants with refractory mantle cell lymphoma (R/R-MCL) who have commenced treatment with lenalidomide after 08 July 2016 (date marketing authorization was granted). Three datasets will be described for the study population and will form the basis of subsequent analyses: Population dataset, Treatment dataset, Outcomes dataset
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
To quantify and characterize the event of TFR by tumor burden in R/R MCL patients treated with lenalidomide in a real-world setting. | Approximately 8.5 years
  To quantify and characterize the event of TFR by tumor burden (assessed based on the last CT scan performed within a maximum of 2 months prior to initiation of administration of lenalidomide) in R/R MCL patients treated with lenalidomide in a real-world setting.

SECONDARY OUTCOMES:
To quantify and characterize the proportion of early deaths by tumor burden in R/R MCL patients treated with lenalidomide in a real-world setting | Approximately 8.5 years
  To quantify and characterize the proportion of early deaths (defined as deaths within 20 weeks of initial administration of lenalidomide) by tumor burden in R/R MCL patients treated with lenalidomide in a real-world setting.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (79):
- Austria (10):
  - Local Institution - 105, Graz
  - LKH Graz Medizinische Universitätsklinik, Graz
  - LKH Hochsteiermark, Standort Leoben, Leoben
  - Local Institution - 104, Leoben
  - Local Institution - 102, Salzburg
  - Salzburger Landeskliniken - Universitaetsklinikum Salzburg, Salzburger
  - AKH Wien, Universitaetsklinik fuer Innere Medizin III, Vienna
  - Local Institution - 101, Vienna
  - Landesklinikum Wiener Neustadt, Wiener Neustadt
  - Local Institution - 103, Wiener Neustadt
- France (8):
  - Centre Hospitalier de Versailles André Mignot, Le Chesnay
  - Local Institution - 303, Le Chesnay
  - Institution: Hopital Prive du Confluent, Nantes
  - Local Institution - 308, Nantes
  - Assistance Publique - Hopitaux de Paris (AP-HP) - Hopital Universitaire Pitie Salpetriere (Hopital Pitie-Salpetriere), Paris
  - Centre Hospitalier de Saint-Quentin, Saint Quentin Picardie
  - Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse
  - Local Institution - 305, Toulouse
- Germany (4):
  - Berufsausuebungsgemeinschaft Kiehl/Stein, Frankfurt/ Oder Brandenburg
  - Praxis fuer Haematolgie, Onkologie und Palliativmedizin, Leipzig
  - Local Institution - 256, Würzburg
  - Universitaetsklinikum Wuerzburg, Würzburg
- Greece (11):
  - General University Hospital of Alexandroupolis, Alexandrouppoli
  - General Anti-Cancer Hospital "Agios Savvas", Athens
  - Local Institution - 501, Athens
  - Private hospital "Iatriko Psychikou", Athens, Athens
  - General University Hospital of Athens "LAIKO", Athens, Athens
  - Local Institution - 502, Athens
  - Local Institution - 506, Athens Goudi
  - General University Hospital "Attikon", Chaïdári
  - Metaxa Cancer Hospital, Athens, Piraeous
  - Local Institution - 511, Rio, Patras
  - Theageneio General Hospital, Thessaloniki, Thessaloniki
- Italy (31):
  - Local Institution - 601, Busto Arsizio
  - Ospedale di Busto Arsizio - ASST Valle Olona, Busto Arsizio
  - Local Institution - 607, Genova
  - Ospedale Policlinico San Martino - IRCCS, Genova
  - Istituto Clinico Humanitas IRCCS, Milan
  - Fondazione IRCCS Ca' Cranda, Ospedale Maggiore Policinico, Milan
  - Local Institution - 614, Milan
  - Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliera Niguarda Ca' Granda, Milan
  - Local Institution - 603, Milan
  - Local Institution - 617, Padua
  - Azienda Ospedaliera di Padova - U.O.C. di Gastroenterologia, Padua
  - Local Institution - 613, Padua
  - Azienda Ospedaliero - Universiaria di Parma, Parma
  - Amyloidosis Research & Treatment Center, Fondazione Irccs Policlinico San Matteo, Pavia
  - Local Institution - 609, Pavia
  - Local Institution - 610, Pisa
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Arcispedale Santa Maria Nuova - AUSL Reggio Emilia, Reggio Emilia
  - Local Institution - 602, Reggio Emilia
  - Infermi Hospital, Rimini
  - Local Institution - 605, Rimini
  - Policlinico Umberto I , Universita La Sapienza, Roma
  - Local Institution - 611, Rome
  - Local Institution - 608, Siena
  - Universita di Siena -Azienda Ospedaliera Universitaria Senese-Policlincio Santa Maria Alle Scotte, Siena
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Torino
  - Local Institution - 616, Torino
  - Presidio Ospedaliero Molinette - A.O.U. Citta della Salute e della Scieza, Torino
  - Ospedale Dell'Angelo Di Mestre, Venezia
  - Local Institution - 606, Venezia - Mestre
- Netherlands (2):
  - HagaZiekenhuis van Den Haag - Juliana Kinderziekenhuis (JKZ) - Leyweg, The Hague
  - Local Institution - 401, The Hague
- Spain (13):
  - Local Institution - 204, Alava
  - Hospital universitario de Alava, Alava País Vasco
  - Hospital Universitario 12 de Octubre, Madrid
  - Local Institution - 207, Madrid
  - Local Institution - 201, Málaga
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital de Orense, Ourense
  - Local Institution - 206, Ourense
  - Local Institution - 202, Salamanca
  - Hospital Clínico Universiatrio de Salamanca, Salamanca
  - Local Institution - 209, Santa Cruz de Tenerife
  - Local Institution - 205, Seville
  - Nuestra Senora de Valme, Seville